CLINICAL TRIAL: NCT00711269
Title: Randomized, Placebo-controlled, Double-blind, Parallel-group, Confirmatory Study of SM-13496 (Lurasidone HCl) in Patients With Schizophrenia <Phase III Study>
Brief Title: Study of SM-13496 (Lurasidone HCl) in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1001002; JapicCTI-080585 (Registry Identifier: JAPIC Clinical Trials Information)
Record Dates: First submitted 2008-06-11; First posted 2008-07-08 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride; Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- SM-13496 (lurasidone HCl) 40mg (Experimental): SM-13496 40 mg was administered orally once daily.
  Interventions: Drug: SM-13496 (lurasidone HCl)
- SM-13496 (lurasidone HCl) 80mg (Experimental): SM-13496 80mg was administered orally once daily.
  Interventions: Drug: SM-13496 (lurasidone HCl)
- Placebo (Placebo Comparator): Placebo was administered orally twice daily.
  Interventions: Drug: Placebo
- Risperidone (Active Comparator): Risperidone was administered orally twice daily.
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: SM-13496 (lurasidone HCl) — Lurasidone HCl: 40 mg/day
  Arms: SM-13496 (lurasidone HCl) 40mg
Drug: SM-13496 (lurasidone HCl) — Lurasidone HCl: 80 mg/day
  Arms: SM-13496 (lurasidone HCl) 80mg
Drug: Placebo
  Arms: Placebo
Drug: Risperidone
  Arms: Risperidone

SUMMARY:
The study evaluates the efficacy and safety of SM-13496 compared with placebo in patients with schizophrenia.

ELIGIBILITY:
Main Inclusion Criteria:

* Patient meets DSM-IV criteria for schizophrenia.
* Patient is 18 or older but younger than 75 years of age on the day of signing informed consent.
* Patient understands the objectives, nature, and other aspects of the study and voluntarily agrees to participate in the study by providing written informed consent.

Main Exclusion Criteria:

* Patient has a history of neuroleptic malignant syndrome, water intoxication, or paralytic ileus.
* Patient has Parkinson's disease.
* Patient has a history or complication of malignancy.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2008-06-27 (Actual); Primary Completion 2010-04-27 (Actual); Study Completion 2010-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Drug Development Division, Study Director — Sumitomo Pharma Co., Ltd.
Locations (3):
- Japan: 67 sites, Tokyo, Etc., Japan
- Korea: 14 sites, Seoul, Etc., South Korea
- Taiwan: 11 sites, Taipei, Etc., Taiwan

RESULTS

PARTICIPANT FLOW:
Groups:
- SM-13496 (Lurasidone HCl) 40-mg Group: SM-13496 40 mg was administered orally once daily.
- SM-13496 (Lurasidone HCl) 80-mg Group: SM-13496 80 mg was administered orally once daily.
- Placebo Group: Placebo was administered orally twice daily.
- Risperidone Group: Risperidone was administered orally twice daily.
Period: Overall Study
Arm/Group | SM-13496 (Lurasidone HCl) 40-mg Group | SM-13496 (Lurasidone HCl) 80-mg Group | Placebo Group | Risperidone Group
Started | 131 | 131 | 133 | 65
Completed | 87 | 83 | 83 | 51
Not Completed | 44 | 48 | 50 | 14

BASELINE CHARACTERISTICS:
Groups:
- Risperidone Group: Risperidone 2 mg was administered orally twice daily.
- Total: Total of all reporting groups
Arm/Group | SM-13496 (Lurasidone HCl) 40-mg Group | SM-13496 (Lurasidone HCl) 80-mg Group | Placebo Group | Risperidone Group | Total
Number analyzed (Participants) | 125 | 129 | 129 | 64 | 447
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (14.48) | 45.7 (13.51) | 46.0 (12.85) | 44.8 (12.59) | 45.6 (13.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 47 | 57 | 29 | 183
  Male | 75 | 82 | 72 | 35 | 264
Region of Enrollment [Number; unit: participants]
  Japan | 63 | 64 | 61 | 33 | 221
  Taiwan | 34 | 37 | 38 | 16 | 125
  Korea, Republic of | 28 | 28 | 30 | 15 | 101

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Positive and Negative Syndrome Scale (PANSS) Total Score at Week 6 (LOCF)
Description: The PANSS is an interview-based measure of the severity of psychopathology in adults with psychotic disorders. The measure is comprised of 30 items and three subscales: the Positive subscale contains seven questions to assess delusions, conceptual disorganization, hallucinations behavior, excitement, grandiosity, suspiciousness/persecution, and hostility; the Negative subscale contains seven questions to assess blunted effect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, lack of motivation, and similar symptoms; and the General Psychopathology subscale addresses other symptoms such as anxiety, somatic concern, and disorientation. An anchored Likert scale from 1-7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. The PANSS total score is the sum of all 30 items and ranges from 30 through 210. A higher score is associated with greater illness severity.
Time Frame: Baseline and Week 6 [Last Observation Carried Forward (LOCF)]
Population: FAS (Full Analysis Set)
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | SM-13496 (Lurasidone HCl) 40-mg Group | SM-13496 (Lurasidone HCl) 80-mg Group | Placebo Group | Risperidone Group
Number analyzed (Participants) | 125 | 129 | 129 | 64
units on a scale | -6.1 (1.75) | -4.3 (1.72) | -2.5 (1.72) | -7.1 (2.44)
Statistical Analysis 1: Comparison: SM-13496 (Lurasidone HCl) 40-mg Group vs Placebo Group; Test type: Superiority — One-way Analysis of Variance (ANOVA); p = 0.149, ANOVA; LS Mean difference = -3.5, 95% CI 2-sided [-8.4 to 1.3] — [Not specified]
Statistical Analysis 2: Comparison: SM-13496 (Lurasidone HCl) 80-mg Group vs Placebo Group; Test type: Superiority — One-way Analysis of variance (ANOVA); p = 0.462, ANOVA; LS Mean difference = -1.8, 95% CI 2-sided [-6.6 to 3.0]
Statistical Analysis 3: Comparison: Placebo Group vs Risperidone Group; Test type: Superiority — One-way Analysis of variance (ANOVA); p = 0.122, ANOVA; LS Mean difference = -4.6, 95% CI 2-sided [-10.5 to 1.2]
Statistical Analysis 4: Comparison: SM-13496 (Lurasidone HCl) 40-mg Group vs SM-13496 (Lurasidone HCl) 80-mg Group vs Placebo Group; Test type: Superiority — Maximum Contrast Method; p = 0.235, Maximum Contrast Method — Contrast Factors (Placebo, SM-13496 40-mg, SM-13496 80-mg): (-1, 0, 1) Adjusted P Value: 0.298; Contrast (Placebo, SM-13496 40-mg, SM-13496 80-mg):(-2, 1, 1) Raw P Value: 0.108 Adjusted P Value: 0.145

2. Secondary Outcome: Change From Baseline in the PANSS Positive Subscales at Week 6 (LOCF)
Description: The PANSS is comprised of 30 items and three subscales. The Positive subscale contains seven questions to assess delusions, conceptual disorganization, hallucinations behavior, excitement, grandiosity, suspiciousness/persecution, and hostility. An anchored Likert scale from 1-7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. The PANSS Positive subscale score is the sum of all 7 items and ranges from 7 through 49. A higher score is associated with greater illness severity.
Time Frame: Baseline and Week 6 (LOCF)
Population: FAS (Full Analysis Set)
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | SM-13496 (Lurasidone HCl) 40-mg Group | SM-13496 (Lurasidone HCl) 80-mg Group | Placebo Group | Risperidone Group
Number analyzed (Participants) | 125 | 129 | 129 | 64
units on a scale | -2.0 (0.55) | -1.4 (0.54) | -0.6 (0.54) | -2.9 (0.77)
Statistical Analysis 1: Comparison: SM-13496 (Lurasidone HCl) 40-mg Group vs Placebo Group; Test type: Superiority — One-way Analysis of variance (ANOVA); p = 0.069, ANOVA; LS Mean difference = -1.4, 95% CI 2-sided [-2.9 to 0.1]
Statistical Analysis 2: Comparison: SM-13496 (Lurasidone HCl) 80-mg Group vs Placebo Group; Test type: Superiority — One-way Analysis of variance (ANOVA); p = 0.287, ANOVA; LS Mean difference = -0.8, 95% CI 2-sided [-2.3 to 0.7]
Statistical Analysis 3: Comparison: Placebo Group vs Risperidone Group; Test type: Superiority — One-way Analysis of variance (ANOVA); p = 0.016, ANOVA; LS Mean difference = -2.3, 95% CI 2-sided [-4.1 to -0.4]

3. Secondary Outcome: Change From Baseline in the PANSS Negative Subscales at Week 6
Description: The PANSS is comprised of 30 items and three subscales. The Negative subscale contains seven questions to assess blunted effect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, lack of motivation, and similar symptoms. An anchored Likert scale from 1-7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. The PANSS Negative subscale score is the sum of all 7 items and ranges from 7 through 49. A higher score is associated with greater illness severity.
Time Frame: Baseline and Week 6 (LOCF)
Population: FAS (Full Analysis Set)
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | SM-13496 (Lurasidone HCl) 40-mg Group | SM-13496 (Lurasidone HCl) 80-mg Group | Placebo Group | Risperidone Group
Number analyzed (Participants) | 125 | 129 | 129 | 64
units on a scale | -1.6 (0.47) | -1.7 (0.46) | -0.9 (0.46) | -1.7 (0.65)
Statistical Analysis 1: Comparison: SM-13496 (Lurasidone HCl) 40-mg Group vs Placebo Group; Test type: Superiority — One-way Analysis of variance (ANOVA); p = 0.289, ANOVA; LS Mean difference = -0.7, 95% CI 2-sided [-2.0 to 0.6]
Statistical Analysis 2: Comparison: SM-13496 (Lurasidone HCl) 80-mg Group vs Placebo Group; Test type: Superiority — One-way Analysis of variance (ANOVA); p = 0.256, ANOVA; LS Mean difference = -0.7, 95% CI 2-sided [-2.0 to 0.5]
Statistical Analysis 3: Comparison: Placebo Group vs Risperidone Group; Test type: Superiority — One-way Analysis of variance (ANOVA); p = 0.352, ANOVA; LS Mean difference = -0.7, 95% CI 2-sided [-2.3 to 0.8]

4. Secondary Outcome: Change From Baseline in the PANSS General Psychopathology Subscales at Week 6 (LOCF)
Description: The PANSS is comprised of 30 items and three subscales. The General Psychopathology subscale addresses other 16 symptoms such as anxiety, somatic concern, and disorientation. An anchored Likert scale from 1-7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. The PANSS General Psychopathology subscale score is the sum of all 16 items and ranges from 16 through 112. A higher score is associated with greater illness severity.
Time Frame: Baseline and Week 6 (LOCF)
Population: FAS (Full Analysis Set)
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | SM-13496 (Lurasidone HCl) 40-mg Group | SM-13496 (Lurasidone HCl) 80-mg Group | Placebo Group | Risperidone Group
Number analyzed (Participants) | 125 | 129 | 129 | 64
units on a scale | -2.4 (0.90) | -1.2 (0.88) | -1.0 (0.88) | -2.6 (1.25)
Statistical Analysis 1: Comparison: SM-13496 (Lurasidone HCl) 40-mg Group vs Placebo Group; Test type: Superiority — One-way Analysis of variance (ANOVA); p = 0.251, ANOVA; LS Mean difference = -1.4, 95% CI 2-sided [-3.9 to 1.0]
Statistical Analysis 2: Comparison: SM-13496 (Lurasidone HCl) 80-mg Group vs Placebo Group; Test type: Superiority — One-way Analysis of variance (ANOVA); p = 0.847, ANOVA; LS Mean difference = -0.2, 95% CI 2-sided [-2.7 to 2.2]
Statistical Analysis 3: Comparison: Placebo Group vs Risperidone Group; Test type: Superiority — One-way Analysis of variance (ANOVA); p = 0.292, ANOVA; LS Mean difference = -1.6, 95% CI 2-sided [-4.6 to 1.4]

5. Secondary Outcome: Proportion of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Proportion of participants with treatment-emergent adverse events. An adverse event was defined as any untoward medical occurrence in a study participant who was taking a medicinal (investigational) product. Treatment-emergent adverse events (TEAEs) were defined as adverse events with a start date on or after the date of the first dose through the end of follow-up, or adverse events occurring before the date of first dose and worsening during the treatment or follow-up period.
Time Frame: From Baseline to up to 8 weeks
Population: Safety population defined as subjects who receive at least one dose of the study drug in the treatment period.
Measure: Count of Participants; unit: Participants
Groups:
- Risperidone Group: Placebo was administered orally twice daily.
Arm/Group | SM-13496 (Lurasidone HCl) 40-mg Group | SM-13496 (Lurasidone HCl) 80-mg Group | Placebo Group | Risperidone Group
Number analyzed (Participants) | 127 | 131 | 132 | 65
Participants | 105 | 103 | 101 | 53

6. Secondary Outcome: Proportion of Participants With TEAEs Leading to Discontinuation
Time Frame: From Baseline to up to 8 weeks
Population: Safety population defined as subjects who receive at least one dose of the study drug in the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | SM-13496 (Lurasidone HCl) 40-mg Group | SM-13496 (Lurasidone HCl) 80-mg Group | Placebo Group | Risperidone Group
Number analyzed (Participants) | 127 | 131 | 132 | 65
Participants | 18 | 18 | 27 | 7

7. Secondary Outcome: Proportion of Participants With Treatment-emergent Serious Adverse Events (SAEs)
Description: Proportion of participants with treatment-emergent adverse events. An adverse event was considered serious if it met one or more of the following criteria: Resulted in death; Was life-threatening (i.e., a patient was at immediate risk of death at the time of the event, not an event where occurrence in a more severe form might have caused death); Required in-patient hospitalization or prolongation of existing hospitalization; Resulted in persistent or significant disability/incapacity; Was a congenital anomaly/birth defect; Was considered to be an important medical event.
Time Frame: From Baseline to up to 8 weeks
Population: Safety population defined as subjects who receive at least one dose of the study drug in the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | SM-13496 (Lurasidone HCl) 40-mg Group | SM-13496 (Lurasidone HCl) 80-mg Group | Placebo Group | Risperidone Group
Number analyzed (Participants) | 127 | 131 | 132 | 65
Participants | 8 | 7 | 10 | 2

ADVERSE EVENTS:
Time Frame: From Baseline to up to 8 weeks
Description: Treatment-emergent adverse events (TEAEs) were defined as adverse events (AEs) with a start date on or after the date of the first dose through the end of follow-up, or AEs occurring before the date of first dose and worsening during the treatment or follow-up period. Both TEAEs and treatment-emergent serious AEs are presented for the safety population defined as subjects who receive at least one of the study drug in the treatment phase.
Groups:
- SM-13496 (Lurasidone HCl) 40-mg Group: SM-13496 40 mg was administered orally once daily, for 6 weeks.
- SM-13496 (Lurasidone HCl) 80-mg Group: SM-13496 40 mg was administered orally once daily on Days 1 to 7, SM-13496 60 mg on Days 8 to 14, and SM-13496 80 mg on Days 15 to 42.
- Placebo Group: Placebo was administered orally twice daily for 6 weeks.
- Risperidone Group: Risperidone 2 mg was administered orally twice daily on Days 1 to 7, risperidone 3 mg on Days 8 to 14, and risperidone 4 mg on Days 15 to 42.
Arm/Group | SM-13496 (Lurasidone HCl) 40-mg Group | SM-13496 (Lurasidone HCl) 80-mg Group | Placebo Group | Risperidone Group
All-Cause Mortality (participants affected / at risk) | 0/127 | 1/131 | 0/132 | 0/65
Serious Adverse Events (participants affected / at risk) | 8/127 | 7/131 | 10/132 | 2/65
Other Adverse Events (participants affected / at risk) | 97/127 | 124/131 | 91/132 | 51/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SM-13496 (Lurasidone HCl) 40-mg Group (N=127) | SM-13496 (Lurasidone HCl) 80-mg Group (N=131) | Placebo Group (N=132) | Risperidone Group (N=65)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0
Nausea (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0
Sudden death (General disorders) | 0 | 1 (1) | 0 | 0
Cellulitis (Infections and infestations) | 1 (1) | 0 | 1 (1) | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 (1) | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 (1) | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0
Convulsion (Nervous system disorders) | 0 | 1 (1) | 0 | 0
Neuroleptic malignant syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 (1)
Schizophrenia (Psychiatric disorders) | 3 (3) | 2 (2) | 6 (6) | 0
Psychotic disorder (Psychiatric disorders) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SM-13496 (Lurasidone HCl) 40-mg Group (N=127) | SM-13496 (Lurasidone HCl) 80-mg Group (N=131) | Placebo Group (N=132) | Risperidone Group (N=65)
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1
Dermoid cyst (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 2 | 1 | 0 | 0
Asthenopia (Eye disorders) | 1 | 0 | 1 | 0
Oculogyric crisis (Eye disorders) | 0 | 1 | 1 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 11 | 13 | 11 | 4
Constipation (Gastrointestinal disorders) | 10 | 11 | 14 | 12
Nausea (Gastrointestinal disorders) | 9 | 4 | 6 | 2
Diarrhoea (Gastrointestinal disorders) | 8 | 4 | 9 | 2
Dyspepsia (Gastrointestinal disorders) | 5 | 3 | 4 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 3 | 4 | 3 | 3
Toothache (Gastrointestinal disorders) | 4 | 1 | 6 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Gingivitis (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 3 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Periodontitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 4 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chapped lips (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Faecal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 2 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Breath odour (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oesophageal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 4 | 5 | 1
Malaise (General disorders) | 1 | 2 | 0 | 0
Oedema peripheral (General disorders) | 2 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Irritability (General disorders) | 0 | 1 | 0 | 0
Thirst (General disorders) | 0 | 1 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 1
Secretion discharge (General disorders) | 0 | 0 | 1 | 0
Allergy to arthropod sting (Immune system disorders) | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 13 | 13 | 13 | 9
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 1 | 3
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Adenoviral conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Carbuncle (Infections and infestations) | 0 | 1 | 0 | 0
Eyelid infection (Infections and infestations) | 0 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0
Purulence (Infections and infestations) | 1 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 1
Dermatitis infected (Infections and infestations) | 0 | 0 | 1 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 2 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Excoriation (Injury, poisoning and procedural complications) | 4 | 4 | 2 | 2
Contusion (Injury, poisoning and procedural complications) | 4 | 1 | 3 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Device breakage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Mouth injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Nail avulsion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 3
Foreign body trauma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Urethral injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 4 | 2 | 2 | 0
Weight increased (Investigations) | 2 | 2 | 1 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 2 | 0 | 0
Weight decreased (Investigations) | 2 | 1 | 5 | 0
Blood pressure decreased (Investigations) | 2 | 0 | 0 | 1
Blood pressure increased (Investigations) | 1 | 1 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 1 | 1 | 0
Protein urine present (Investigations) | 1 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 1 | 0
Blood prolactin increased (Investigations) | 1 | 0 | 0 | 5
Blood uric acid increased (Investigations) | 1 | 0 | 0 | 1
Glucose urine present (Investigations) | 0 | 1 | 0 | 0
Platelet count increased (Investigations) | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 1 | 0
Deoxypyridinoline urine increased (Investigations) | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 6 | 3 | 2 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Oral intake reduced (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 4 | 3 | 4 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Akathisia (Nervous system disorders) | 11 | 15 | 6 | 9
Headache (Nervous system disorders) | 8 | 11 | 10 | 3
Tremor (Nervous system disorders) | 3 | 10 | 8 | 5
Somnolence (Nervous system disorders) | 4 | 6 | 2 | 0
Dyskinesia (Nervous system disorders) | 3 | 5 | 4 | 2
Dystonia (Nervous system disorders) | 2 | 6 | 1 | 3
Parkinsonian gait (Nervous system disorders) | 2 | 5 | 0 | 1
Dizziness (Nervous system disorders) | 3 | 3 | 2 | 0
Sedation (Nervous system disorders) | 2 | 3 | 2 | 2
Bradykinesia (Nervous system disorders) | 1 | 2 | 3 | 3
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Autism (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 1
Drooling (Nervous system disorders) | 0 | 0 | 1 | 0
Parkinsonism (Nervous system disorders) | 0 | 0 | 1 | 0
Tardive dyskinesia (Nervous system disorders) | 0 | 0 | 1 | 0
Schizophrenia (Psychiatric disorders) | 15 | 25 | 25 | 10
Insomnia (Psychiatric disorders) | 18 | 25 | 19 | 4
Psychotic disorder (Psychiatric disorders) | 0 | 3 | 3 | 0
Agitation (Psychiatric disorders) | 1 | 3 | 4 | 0
Aggression (Psychiatric disorders) | 0 | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 5 | 2
Depressive symptom (Psychiatric disorders) | 0 | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 1 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 0 | 1 | 0
Dissociative disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 2 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Galactorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Menstruation delayed (Reproductive system and breast disorders) | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 5 | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 3 | 4 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin discomfort (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 1 | 2 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes